CLINICAL TRIAL: NCT00319384
Title: Outpatient Ultrafiltration Therapy in Heart Failure Feasibility Trial
Brief Title: Outpatient Ultrafiltration Therapy in Heart Failure Patients Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: Nuwellis, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR 06-2642
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Congestive Heart Failure
Keywords: congestive heart failure; heart failure; ultrafiltration therapy; fluid overload
MeSH Terms: conditions — Heart Failure; Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Ultrafiltration therapy

SUMMARY:
This trial will look at the effectiveness and patient acceptance of ultrafiltration therapy in an outpatient setting.

The purpose of this study is to determine if ambulatory patients who suffer from heart failure and hypervolemia can be safely and effectively treated in an outpatient infusion clinic. The results from this trial will be useful in planning a larger, randomized trial comparing usual care and ultrafiltration for this patient population in similar ambulatory settings.

DETAILED DESCRIPTION:
This is a pilot study to assess the feasibility, effectiveness, safety and patient acceptance of ultrafiltration in ambulatory patients with heart failure and hypervolemia. The results will be useful in planning a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be recruited from the cardiology clinic at Hennepin County Medical Center. Patients are eligible for the study if they are:

  1. Older than 18
  2. Not pregnant
  3. Have heart failure with worsening hypervolemia despite oral diuretics
  4. Have at least two of the following signs or symptoms of hypervolemia: JVD, edema >1+, rales pulmonary edema on chest x-ray, orthopnea or PND
  5. Not more than 10 kg above their usual baseline weight
  6. Have, in the opinion of the treating physician, a need for a minimum of 2 liters of volume removal

     Exclusion Criteria:

  <!-- -->

  1. Systolic blood pressure < 90 mmHg
  2. Serum creatinine > 3.0 mg/dL
  3. Hematocrit >45 %
  4. Uncontrolled arrhythmias
  5. Need for hospitalization
  6. Require renal replacement therapy
  7. Contraindication to anticoagulation with heparin
  8. Poor venous access.

     -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-04; Study Completion 2007-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy
The primary efficacy endpoint is weight loss measured immediately and 48 hours after ultrafiltration.

SECONDARY OUTCOMES:
Quality of life will be assessed by the NYHA classification at 48 hours.
Likert scales addressing global heart failure and shortness of breath symptoms at 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Bart, MD, Principal Investigator — Hennepin Faculty Associates
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Bart BA, Boyle A, Bank AJ, Anand I, Olivari MT, Kraemer M, Mackedanz S, Sobotka PA, Schollmeyer M, Goldsmith SR. Ultrafiltration versus usual care for hospitalized patients with heart failure: the Relief for Acutely Fluid-Overloaded Patients With Decompensated Congestive Heart Failure (RAPID-CHF) trial. J Am Coll Cardiol. 2005 Dec 6;46(11):2043-6. doi: 10.1016/j.jacc.2005.05.098. Epub 2005 Nov 4. PMID 16325039